CLINICAL TRIAL: NCT05624242
Title: Assessment of Right Ventricular Function by Cardiac Magnetic Resonance Imaging in Patients With Pulmonary Arterial Hypertension (IRMA)
Brief Title: Assessment of Right Ventricular Function by Cardiac MRI in Patients With Pulmonary Arterial Hypertension (IRMA)
Acronym: IRMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI03935
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac magnetic resonance imaging — all patients had magnetic resonance imaging at baseline and during follow-up.

SUMMARY:
Pulmonary hypertension (PH) is a pathophysiological condition defined by an increase in pulmonary arterial pressure above 20mmHg, which encompasses many very dissimilar conditions. Right ventricular function is the major determinant of survival in these patients. Currently, right ventricular function is estimated by trans-thoracic echocardiography via the measurement of standardised parameters. However, cardiac magnetic resonance imaging is now the reference technique for non-invasive quantification of volumes, mass, function of the right ventricle but can also be useful for the consideration of the pulmonary circulation. Thus, indices of function can be extracted and it plays an increasing role in the prognostic evaluation of the right heart function at diagnosis and at re-evaluation under treatment of pulmonary arterial hypertension. This work will initially focus on the assessment of right ventricular myocardial work by echocardiography and cardiac magnetic resonance imaging in comparison with invasive haemodynamic data.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pulmonary arterial hypertension (group 1)
* Patient with cardiac MRI, echocardiography and right heart catheterisation within 1 month of each other

Exclusion Criteria:

* Patient with features of venous/capillary involvement
* Pulmonary arterial hypertension associated with with congenital heart disease
* Patient's decline to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population concerns patients with pulmonary arterial hypertension followed up in our centre, at diagnosis and when starting vasodilator treatment.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Transplantation-free survival | 12 months

IPD SHARING:
Plan to Share IPD: No